CLINICAL TRIAL: NCT02605109
Title: Analysis of Human to Human Transmission of Middle East Respiratory Syndrom Coronavirus (MER-CoV) and Infection Control Experiences in a Medical Institution of South Korea
Brief Title: Analysis of Human to Human Transmission of Middle East Respiratory Syndrom Coronavirus (MER-CoV)
Acronym: MKU
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Assistant Professor, Konkuk University Medical Center
Other Study IDs: MERSKORKUH
Record Dates: First submitted 2015-11-11; First posted 2015-11-16 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Viral Infection
Keywords: MERS-CoV; Infection control; Case-control studies
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RiskMERS: Exposed to case-patients
  Interventions: Other: Risk of MERS infection

INTERVENTIONS:
Other: Risk of MERS infection — HCPs, patients and layperson to closely or indirectly contact a case-patients

SUMMARY:
This study aimed to analysis the characteristics of MERS transmission and the effect of our institutional personal protective equipment on the controlling the MERS at a tertiary Korean Hospital.

DETAILED DESCRIPTION:
Between May 2015 and Nov 2015, total 186 cases of MERS-Cov infections were reported in South Korea. In June 2015, a female patient visited our emergency department (ED) for care of femur fracture. She was suspected of having MERS-Cov and isolated after 10 hours from the visit of our hospital because her clinical feature was not concordance with typical MERS-Cov infection and she denied the any contact of MERS-Cov patient. Before the transport to the isolation room, she stayed at ED during 8 hours, and admitted the general ward during 2 hours. Approximately 150 including the healthcare providers, patients and laypersons were exposed to the case-patient directly or indirectly. The investigators monitored all possible contacts in the hospital during that time, and analysed the CCTV data of hospital and interviewed all risk-persons. After the hospital outbreak ended, The investigators analysed the data of all behavior and contact history of MERS patient, epidermic and clinical data of infected patients and data of personal protective equipments (PPE) of all exposed persons.

Descriptive analysis were conducted for basic epidemiology, transmission rout of MERS in hospital, and the effect of hospital infection control system and PPE of each contacts.

ELIGIBILITY:
Inclusion Criteria:

* All aged persons who have risk of MERS transmission from a case-patients

Exclusion Criteria:

* No risk of transmission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pesons who had the risk of MERS transmission from the case-patient
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Numbers of infected patient | Serologic confimred MERS case within 4 weeks after contacting to a case patients

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kyun Ki, MD, Study Director — Devision of Infection, Department of Medicine, School of Medicine, Konkuk University, Seoul 143-729, Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cetra A. MERS-CoV update: what you need to know. Lancet Infect Dis. 2014 Oct;14(10):924-5. doi: 10.1016/s1473-3099(14)70930-2. No abstract available. PMID 25379596
- [Background] Oh MD, Choe PG, Oh HS, Park WB, Lee SM, Park J, Lee SK, Song JS, Kim NJ. Middle East Respiratory Syndrome Coronavirus Superspreading Event Involving 81 Persons, Korea 2015. J Korean Med Sci. 2015 Nov;30(11):1701-5. doi: 10.3346/jkms.2015.30.11.1701. Epub 2015 Oct 16. PMID 26539018
- [Background] Yang JS, Park S, Kim YJ, Kang HJ, Kim H, Han YW, Lee HS, Kim DW, Kim AR, Heo DR, Kim JA, Kim SJ, Nam JG, Jung HD, Cheong HM, Kim K, Lee JS, Kim SS. Middle East Respiratory Syndrome in 3 Persons, South Korea, 2015. Emerg Infect Dis. 2015 Nov;21(11):2084-7. doi: 10.3201/eid2111.151016. PMID 26488745
- [Background] Korean Society of Infectious Diseases; Korean Society for Healthcare-associated Infection Control and Prevention. An Unexpected Outbreak of Middle East Respiratory Syndrome Coronavirus Infection in the Republic of Korea, 2015. Infect Chemother. 2015 Jun;47(2):120-2. doi: 10.3947/ic.2015.47.2.120. Epub 2015 Jun 30. PMID 26157591
- [Background] Gostin LO, Lucey D. Middle East Respiratory Syndrome: A Global Health Challenge. JAMA. 2015 Aug 25;314(8):771-2. doi: 10.1001/jama.2015.7646. No abstract available. PMID 26084030
- [Background] Zumla A, Hui DS, Perlman S. Middle East respiratory syndrome. Lancet. 2015 Sep 5;386(9997):995-1007. doi: 10.1016/S0140-6736(15)60454-8. Epub 2015 Jun 3. PMID 26049252
- [Result] Kayali G, Peiris M. A more detailed picture of the epidemiology of Middle East respiratory syndrome coronavirus. Lancet Infect Dis. 2015 May;15(5):495-7. doi: 10.1016/S1473-3099(15)70128-3. Epub 2015 Apr 8. No abstract available. PMID 25863563
- [Derived] Ki HK, Han SK, Son JS, Park SO. Risk of transmission via medical employees and importance of routine infection-prevention policy in a nosocomial outbreak of Middle East respiratory syndrome (MERS): a descriptive analysis from a tertiary care hospital in South Korea. BMC Pulm Med. 2019 Oct 30;19(1):190. doi: 10.1186/s12890-019-0940-5. PMID 31666061